CLINICAL TRIAL: NCT05463705
Title: Addressing Diffusion of Responsibility and Prescribing Burden to Improve Use of Diabetes Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nancy Haff, MD, MPH, Associate Epidemiologist, Division of Pharmacoepidemiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022P001663; 5P30AG064199-02 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-07-19 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Diabetes; SGLT-2i and GLP-1RA Therapies; Diffusion of Responsibility; Prescribing Burden
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention to address diffusion of responsibility (Experimental): PCPs will receive an email from a peer offering encouragement and support in prescribing SGLT-2is and GLP-1RAs that includes specific components designed to reduce diffusion of responsibility. Specifically, these elements will be adapted from interventions that mitigate diffusion of responsibility in other contexts, including: (1) assigning responsibility to individuals or smaller groups, (2) increased perceived harm of the situation to be addressed (3) highlighting competence to act, and (4) modeling the desired behavior. The email will also contain a link to clinical and administrative information to support prescribing and an offer for direct support from the peer.
  Interventions: Behavioral: Intervention to address diffusion of responsibility
- Intervention to address diffusion of responsibility + simplification of prescribing (Experimental): PCPs will receive the same contact addressing diffusion of responsibility as in the "Intervention to address diffusion of responsibility" arm, but will additionally have access to an experienced administrative team for diabetes medication insurance authorization support, by "routing" their clinic note through the EHR. PCPs will be informed, suing the same email outreach, how to access the administrative team, which consists of medical and administrative assistants and currently supports prescribing within the endocrinology division. The team will follow up with the pharmacy to determine coverage, complete prior authorizations, determine alternate covered options, and track progress.
  Interventions: Behavioral: Intervention to address diffusion of responsibility + simplification of prescribing
- Usual care (No Intervention): PCPs in this arm will receive no additional outreach or resources than standard MGH primary care practice.

INTERVENTIONS:
Behavioral: Intervention to address diffusion of responsibility — PCPs will receive an email from a peer offering encouragement and support in prescribing SGLT-2is and GLP-1RAs that includes specific components designed to reduce diffusion of responsibility. Specifically, these elements will be adapted from interventions that mitigate diffusion of responsibility in other contexts, including: (1) assigning responsibility to individuals or smaller groups, (2) increased perceived harm of the situation to be addressed (3) highlighting competence to act, and (4) modeling the desired behavior. The email will also contain a link to clinical and administrative information to support prescribing and an offer for direct support from the peer.
  Arms: Intervention to address diffusion of responsibility
Behavioral: Intervention to address diffusion of responsibility + simplification of prescribing — PCPs will receive the same contact addressing diffusion of responsibility as in the "Intervention to address diffusion of responsibility" arm, but will additionally have access to an experienced administrative team for diabetes medication insurance authorization support, by "routing" their clinic note through the EHR. PCPs will be informed, suing the same email outreach, how to access the administrative team, which consists of medical and administrative assistants and currently supports prescribing within the endocrinology division. The team will follow up with the pharmacy to determine coverage, complete prior authorizations, determine alternate covered options, and track progress.
  Arms: Intervention to address diffusion of responsibility + simplification of prescribing

SUMMARY:
This study will test the impact of addressing diffusion of responsibility with and without additional reduction of prescribing burden on SGLT-2i and GLP-1RAs prescribing compared to usual care.

Population: MGH primary care physicians caring for at least 2 eligible patients. Eligible patients are individuals age18 years or older with type 2 diabetes and HbA1c >7.5% and a compelling indication for an SGLT-2i or GLP-1RA (including cardiovascular disease, kidney disease, heart failure, or obesity), who are not already prescribed one of these therapies.

Intervention: PCPs will be randomized to one of three arms: 1) intervention to address diffusion of responsibility, 2) Intervention to address diffusion of responsibility with additional simplification of prescribing, 3) usual care.

DETAILED DESCRIPTION:
This study will be conducted within MGH primary care. As with prior work, the investigators will use the hospital's EHR database, the Epic Enterprise Data Warehouse, to identify patients. Patients will be eligible if they are: adults 18-84 years of age with poorly controlled type 2 diabetes (defined as HbA1c >7.5% for ages 18-69 and >8.5% for ages 70-84) and a compelling indication for an SGLT-2i or GLP-1RA (including cardiovascular disease, kidney disease, heart failure, or obesity), who are not already prescribed one of these therapies. The investigators will exclude individuals with end stage renal disease, dementia, type I diabetes, or an EHR indicator of hospice care. The investigators will also exclude patients who are not on the MGH diabetes registry, because patients who are excluded from the registry typically have a clinical reason for alternative diabetes goals or care plans. PCPs caring for at least one eligible patient will be included in the trial. Eligible PCPs will be randomized to one of three arms: (1) intervention to address diffusion of responsibility, (2) intervention to address diffusion of responsibility plus additional simplification of the prescribing process, and (3) usual care. Providers randomized to arm 1, the intervention to address diffusion of responsibility will receive an email from a peer offering encouragement and support in prescribing SGLT-2is and GLP-1RAs that includes specific components designed to reduce diffusion of responsibility. The email will also contain a link to clinical and administrative information to support prescribing and an offer for direct support from the peer. Providers randomized to arm 2, the intervention addressing diffusion of responsibility and simplifying the prescribing process will receive the same contact addressing diffusion of responsibility as in arm 1, but they will additionally have access to an experienced administrative team for diabetes medication insurance authorization support. The primary outcome will be the rate of prescriptions for SGLT-2is and GLP-1RAs among eligible patients.

ELIGIBILITY:
Inclusion Criteria:

Patients:

We will use EHR data to identify patients

* 18-84 years of age
* Diagnosed with type 2 diabetes
* Has poorly controlled diabetes (defined as HbA1c >7.5% for ages 18-69 and >8.5% for ages 70-84)
* Have a compelling indication for an SGLT-2i or GLP-1RA who are not already prescribed one of these therapies. A compelling indication includes individuals with cardiovascular disease, kidney disease, heart failure, or obesity.

Physicians:

Physicians will be included if they are

* Practicing in primary care at Massachusetts General Hospital
* Caring for at least 1 patient: (1) age 18-84, (2) diagnosed with type 2 diabetes, (3) has poorly controlled diabetes (defined as HbA1c >7.5% for ages 18-69 and >8.5% for ages 70-84) (4) has a compelling indication for an SGLT-2i or GLP-1RA (including cardiovascular disease, kidney disease, heart failure, or obesity), who are not already prescribed one of these therapies.

Exclusion Criteria:

Patients:

* We will exclude individuals with end stage renal disease, dementia, type I diabetes, or an EHR indicator of hospice care.
* We will also exclude patients who are not on the MGH diabetes registry, because patients who are excluded from the registry typically have a clinical reason for alternative diabetes goals or care plans.

Physicians:

- Providers will be excluded if they are involved in the design or conduct of this study (e.g. Drs. Haff and Horn, and the peer PCPs delivering the study intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1580 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haff N, Horn DM, Bhatkhande G, Sung M, Colling C, Wood W, Robertson T, Gaposchkin D, Simmons L, Yang J, Yeh J, Crum KL, Hanken KE, Lauffenburger JC, Choudhry NK. Encouraging the prescribing of SGLT2i and GLP-1RA medications to reduce cardiovascular and renal risk in patients with type 2 diabetes: Rationale and design of a randomized controlled trial. Am Heart J. 2025 Jul;285:39-51. doi: 10.1016/j.ahj.2025.02.007. Epub 2025 Feb 20. PMID 39986337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All primary care physicians at Mass General Hospital who were not participating in the delivery of the study and whose clinics agreed to participation were randomized to study arms.
Pre-assignment Details: All primary care physicians at Mass General Hospital who were not participating in the delivery of the study and whose clinics agreed to participation were randomized to study arms. Eligible patients were identified using routinely-collected electronic health record data and were included in the study if they met inclusion criteria and had an upcoming visit scheduled with their PCP during the intervention period.
Groups:
- Usual Care - Patients; Usual Care - Providers: PCPs in this arm received no additional outreach or resources.
- Intervention to Address Diffusion of Responsibility - Patients: Patients were not intervened upon directly. In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing, electronic health record (EHR) messages containing prescribing tips sent before visits with eligible patients, and a hand-signed note with a prescribing tips sheet from the peer champion.
- Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Patients: Patients were not intervened upon directly. In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing and a hand-signed note with a prescribing tips sheet from the peer champion. In this arm, electronic health record (EHR) messages sent before visits with eligible patients contained information on insurance coverage for SGLT2i and GLP-1RA medications specific to each patient.
- Intervention to Address Diffusion of Responsibility - Providers: In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing, electronic health record (EHR) messages containing prescribing tips sent before visits with eligible patients, and a hand-signed note with a prescribing tips sheet from the peer champion.
- Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Providers: In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing and a hand-signed note with a prescribing tips sheet from the peer champion. In this arm, electronic health record (EHR) messages sent before visits with eligible patients contained information on insurance coverage for SGLT2i and GLP-1RA medications specific to each patient.
Period: Overall Study
Arm/Group | Usual Care - Patients | Intervention to Address Diffusion of Responsibility - Patients | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Patients | Usual Care - Providers | Intervention to Address Diffusion of Responsibility - Providers | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Providers
Started | 459 | 484 | 446 | 62 | 66 | 63
Completed (Only eligible patients who attended a visit with their PCP during the intervention period are included in the primary outcome. Providers were also required to have had at least one visit completed with an eligible patient for inclusion in the primary outcome.) | 356 | 377 | 346 | 58 | 58 | 59
Not Completed | 103 | 107 | 100 | 4 | 8 | 4
Not completed — Did not complete a visit during study intervention period | 103 | 107 | 100 | 4 | 8 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the cohort of randomized patients and providers (1389 patients and 191 providers)
Groups:
- Usual Care - Patients: Patients were not intervened upon directly. PCPs in this arm received no additional outreach or resources.
- Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Providers: In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing and a hand-signed note with a prescribing tips sheet from the peer champion. In this arm, electronic health record (EHR) messages sent before visits with eligible patients contained information on insurance coverage for SGLT2i and GLP-1RA medications specific to the patient.
- Total: Total of all reporting groups
Arm/Group | Intervention to Address Diffusion of Responsibility - Patients | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Patients | Usual Care - Patients | Intervention to Address Diffusion of Responsibility - Providers | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Providers | Usual Care - Providers | Total
Number analyzed (Participants) | 484 | 446 | 459 | 66 | 63 | 62 | 1580
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age variable only known and reported for patient subjects. Provider demographic characteristics were not measured.
  years
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    (all) | 66.4 (11.8) | 65.0 (12.6) | 66.4 (11.9) |  |  |  | 66.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex variable only known and reported for patient subjects. Provider demographic characteristics were not measured.
  Participants
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    Female | 235 | 218 | 191 | 0 | 0 | 0 | 644
    Male | 249 | 228 | 268 | 0 | 0 | 0 | 745
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was only known and reported for patient subjects. Provider demographic characteristics were not measured.
  Participants
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    Hispanic or Latino | 78 | 61 | 79 |  |  |  | 218
    Not Hispanic or Latino | 382 | 352 | 354 |  |  |  | 1088
    Unknown or Not Reported | 24 | 33 | 26 |  |  |  | 83
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race variable only known and reported for patient subjects. Provider demographic characteristics were not measured.
  Participants
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    American Indian or Alaska Native | 0 | 4 | 3 |  |  |  | 7
    Asian | 41 | 48 | 38 |  |  |  | 127
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 |  |  |  | 1
    Black or African American | 63 | 55 | 67 |  |  |  | 185
    White | 299 | 277 | 270 |  |  |  | 846
    More than one race | 0 | 0 | 0 |  |  |  | 0
    Unknown or Not Reported | 81 | 62 | 80 |  |  |  | 223
SGLT2 / GLP1 qualifying condition [Count of Participants; unit: Participants] — Population: Qualifying condition was only known and reported for patient subjects. This was not applicable for providers.
  Participants
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    For SGLT2i (CKD, Heart Failure) ONLY | 18 | 30 | 29 |  |  |  | 77
    For GLP-1RA (Obesity, ASCVD) ONLY | 345 | 292 | 323 |  |  |  | 960
    For both SGLT2i and GLP-1RA | 121 | 124 | 107 |  |  |  | 352
Baseline HbA1c (%) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — Population: Baseline HbA1c is only known and reported for patient subjects. Provider clinical characteristics were not measured.
  percentage of glycated hemoglobin
    number analyzed (Participants) | 484 | 446 | 459 | 0 | 0 | 0 | 1389
    (all) | 8.4 (1.5) | 8.4 (1.5) | 8.4 (1.4) |  |  |  | 8.4 (1.5)
Baseline SGLT2 and GLP-1 Prescribing Rate [Mean (Standard Deviation); unit: percentage] — Population: Baseline prescribing rate was only measured for providers. This is the percentage of each providers' patients with diabetes that were already prescribed a SGLT2i or GLP1-RA at baseline.
  percentage
    number analyzed (Participants) | 0 | 0 | 0 | 66 | 63 | 62 | 191
    (all) |  |  |  | 25.4 (10.7) | 25.1 (12.4) | 26.0 (11.8) | 25.5 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prescriptions for SGLT-2i or GLP-1RA Medications Among Eligible Patients in Each Arm
Description: Electronic health record (EHR) prescribing data was used to identify the number of patients with prescriptions for SGLT-2i and GLP-1RA medications beginning 3 business days before the targeted patient visit and continuing through 28 days after the visit. The primary outcome only includes patients who attended the targeted visit.
Time Frame: Beginning 3 days before the targeted visit and continuing through 28 days after the visit
Population: This analysis includes only patients who attended the targeted visit.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention to Address Diffusion of Responsibility: In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing, electronic health record (EHR) messages containing prescribing tips sent before visits with eligible patients, and a hand-signed note with a prescribing tips sheet from the peer champion.
- Intervention to Address Diffusion of Responsibility + Simplification of Prescribing: In this arm, PCPs received support for SGLT2i and GLP-1RA prescribing from the peer champions including a welcome email offering encouragement and support in prescribing and a hand-signed note with a prescribing tips sheet from the peer champion. In this arm, electronic health record (EHR) messages sent before visits with eligible patients contained information on insurance coverage for SGLT2i and GLP-1RA medications specific to each patient.
- Usual Care: PCPs in this arm received no additional outreach or resources.
Arm/Group | Intervention to Address Diffusion of Responsibility | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing | Usual Care
Number analyzed (Participants) | 377 | 346 | 356
Participants | 109 | 92 | 92
Statistical Analysis 1: Comparison: Intervention to Address Diffusion of Responsibility vs Usual Care; Test type: Equivalence — We estimated that 178 providers caring for 1,249 eligible patients would provide 80% power to observe an 11 percentage-point difference in prescribing rates between each intervention arm and control, assuming a control arm prescribing rate of 30%, an ICC of 0.07 (estimated based on prior studies in this system), an average of 7 patients per provider, and a type I error rate of 5%; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.88 to 1.96]
Statistical Analysis 2: Comparison: Intervention to Address Diffusion of Responsibility + Simplification of Prescribing vs Usual Care; Test type: Equivalence — We estimated that 178 providers caring for 1,249 eligible patients would provide 80% power to observe an 11 percentage-point difference in prescribing rates between each intervention arm and control, assuming a control arm prescribing rate of 30%, an ICC of 0.07 (estimated based on prior studies in this system),72,73 an average of 7 patients per provider, and a type I error rate of 5%; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.66 to 1.52]

2. Secondary Outcome: Number of Participants With Prescriptions for SGLT-2i or GLP-1RA Medications Among All Study-eligible Patients, Compared Across Study Arms
Description: Electronic health record (EHR) prescribing data was used to identify patients with prescriptions for SGLT-2i and GLP-1RA medications beginning 3 business days before the targeted patient visit and continuing through 28 days after the visit. This outcome includes all study-eligible patients, regardless of whether they attended the targeted visit.
Time Frame: Beginning 3 days before the targeted visit and continuing through 28 days after the visit
Population: This outcome includes all study-eligible patients, regardless of whether they attended the targeted visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention to Address Diffusion of Responsibility | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing | Usual Care
Number analyzed (Participants) | 484 | 446 | 459
Participants | 134 | 110 | 117
Statistical Analysis 1: Comparison: Intervention to Address Diffusion of Responsibility vs Usual Care; Test type: Superiority — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.83 to 1.61]
Statistical Analysis 2: Comparison: Intervention to Address Diffusion of Responsibility + Simplification of Prescribing vs Usual Care; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.64 to 1.30]

3. Secondary Outcome: Change in Hemoglobin A1c (A1c) Over 6 Months, Compared Across Study Arms
Description: EHR data was used to identify Hemoglobin A1c values. The baseline A1c was the last A1c measured within the 6-months prior to the targeted visit, and the follow-up A1c was the A1c measured between 3 and 9 months after the targeted visit and closest to 6 months after the targeted visit. The change in A1c was calculated and compared across study arms. This analysis includes all patients who had an A1c in follow-up.
Time Frame: 6 months
Population: This analysis includes all patients who had an A1c between 3 and 9 months after the targeted visit.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention to Address Diffusion of Responsibility | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing | Usual Care
Number analyzed (Participants) | 317 | 293 | 295
percentage of glycated hemoglobin | -0.51 (1.44) | -0.51 (1.76) | -0.58 (1.55)
Statistical Analysis 1: Comparison: Intervention to Address Diffusion of Responsibility vs Usual Care; Test type: Superiority; Difference in HbA1c % = 0.18, 95% CI 2-sided [-0.07 to 0.43]
Statistical Analysis 2: Comparison: Intervention to Address Diffusion of Responsibility vs Usual Care; Test type: Superiority; Difference in HbA1c % = 0.06, 95% CI 2-sided [-0.22 to 0.34]

ADVERSE EVENTS:
Time Frame: Adverse events were passively collected for patients. Adverse event monitoring began the day each patient entered the study and continued through the 6-month follow-up period. Additionally, any adverse events that were noted during chart review data collection through the primary completion date were captured and reported.
Description: Because this was a low-risk study conducted within routine primary care, adverse events were monitored passively through information reported to the study team by physician participants as well as through general monitoring of the safety reporting system used within the practices that is reviewed by the study site lead. This monitoring plan was approved by the study's DSMB and reporting was conducted throughout the study.
Arm/Group | Usual Care - Patients | Intervention to Address Diffusion of Responsibility - Patients | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Patients | Usual Care - Providers | Intervention to Address Diffusion of Responsibility - Providers | Intervention to Address Diffusion of Responsibility + Simplification of Prescribing - Providers
All-Cause Mortality (participants affected / at risk) | 3/459 | 1/484 | 2/446 | 0/62 | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/459 | 0/484 | 0/446 | 0/62 | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 0/459 | 0/484 | 0/446 | 0/62 | 0/66 | 0/63

LIMITATIONS AND CAVEATS:
Single site study that already had a high level of SGLT2i and GLP-1RA prescribing at baseline. For some patients medications were not affordable even with guidance on insurance coverage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT05463705/Prot_SAP_000.pdf